CLINICAL TRIAL: NCT02900755
Title: Effects of Perampanel on Cognition and Electroencephalography in Patients With Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Young Jung, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1602-107-742
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Electroencephalography
Keywords: Electroencephalography; Perampanel
MeSH Terms: interventions — perampanel

ARMS (1):
- Epilepsy (Experimental): Epilepsy patients (focal onset seizure with or without secondary generalization)
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — The subjects will be administered oral perampanel for six months. Dose will be titrated according to the tolerance and be maintained at least 1 month before second EEG evaluation.
  Other Names: Fycompa

SUMMARY:
Perampanel, a novel AED, has been recently authorized in Korea and worldwide as a treatment of refractory partial-onset seizures with a new anti-epileptic mechanism of a selective non-competitive antagonist of AMPA receptors.

Evaluating adverse effects during the introduction of new AED is often difficult since the complaints are subjective and objective assessment is complicated due to the polytherapy. Majority of previous studies are focused on quantitative analysis of EEG for taking new AEDs because of the correlation of EEG analysis results and side effects of AED such as cognitive slowing. Therefore, this study aims to investigate the effects of perampanel on EEG in terms of EEG background spectra and to evaluate perampanel effects by using subjective questionnaires assessing depression, anxiety, sleep quality and fatigue.

DETAILED DESCRIPTION:
Perampanel is a selective antagonist of the α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) receptor and is used to treat partial-onset seizures with or without secondary generalization. This antiepileptic drug (AED) is usually prescribed as adjunctive treatment and is also used primarily in generalized tonic-clonic seizures Cognitive dysfunction is a major comorbidity in many patients with epilepsy and could be the result of chronic use of AEDs. Since cognitive decline has a tremendous impact on the quality of life, the effect of a large number of AEDs on cognition has been actively studied. It has been reported that AEDs such as gabapentin, carbamazepine, and topiramate induce cognitive decline, while lamotrigine, levetiracetam, and oxcarbazepine show much less negative effect on cognitive function compared with the older AEDs. Perampanel has also been studied for its effects on cognition in adolescent patients with epilepsy aged 12-18 years. However, the effects of perampanel on cognitive function have not yet been studied in adults.

Electroencephalogram (EEG) spectral analysis or quantitative EEG (QEEG) is a method of quantifying the different frequencies in EEG signals. Spectral analysis of EEG frequency can reflect the functional state of the brain. Thus, it has proved to be a useful tool for assessing the pharmacological effects of central nervous system (CNS) drugs. Electrophysiologic changes due to AEDs can manifest as either a generalized slowing of or an increased beta frequency on EEG in general. Changes in background EEG may be correlated with clinical cognitive function. Since EEG changes in the spectral analysis are only intended to assess brain activity and do not directly reflect clinical changes in patients, neuropsychological (NP) tests are necessary for evaluating clinical cognitive function. Our objective was to determine how perampanel affects cognition and the EEG signal in adult patients with epilepsy. Correlation of these effects was also analyzed with the serum concentration of perampanel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-65 years
* Provide written informed consent signed by the subject or legal guardian prior to entering the study in accordance with the IRB guidelines
* Subjects in otherwise good health (with the exception of epilepsy), as determined by the PI via the medical history, a physical examination and screening laboratory investigations including demonstration of normal renal function.
* Patient with focal-onset seizures with or without secondary generalized seizure
* History of epilepsy for at least 2 years.
* The subject must have had an EEG or clinical seizure consistent with partial epilepsy.

Exclusion Criteria:

* A history of non-epileptic or psychogenic seizures.
* Women who are pregnant or lactating.
* Any clinically significant laboratory abnormality which, in the opinion of the investigator, will exclude the subject from the study.
* Liver transammases (AST and ALT) cannot exceed twice the upper limit of normal and total and direct bilirubin must be within normal limits.
* An active CNS infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
* Any clinically significant psychiatric illness, psychological or behavioral problems which, in the opinion of the investigator, would interfere with the subject's ability to participate in the study.
* Suffering from psychotic disorders and/or unstable recurrent affective disorders evident by use of antipsychotics; subject with current major depressive episode (or within 6 months).
* A history of alcoholism, drug abuse, or drug addiction within the past 2 years.
* History of regular alcohol consumption exceeding 2-3 units/day for females and 3-4 units/day for males
* History of regular use of tobacco or nicotine-containing products exceeding the equivalent of 5 cigarettes per day
* History of regular consumption of caffeine exceeding the equivalent of 4 cups of coffee per day, a level that approximates health-related criteria
* Subject has had greater than 2 allergic reactions to an AED or one serious hypersensitivity reaction to an AED.
* Subjects with more than 1 lifetime suicide attempt or any suicide attempt within the past two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2019-04 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Quantitative EEG (qEEG) change | 6th month
  Change of qEEG markers
  - spectral power: delta, theta, alpha and beta frequency band

SECONDARY OUTCOMES:
Effects on cognition | 6th month
  global cognitive function: Mini-mental state examination Attention and working memory: Digit span forward and backward Frontal/Executive function: Stroop test, trail-making test (TMT, A -and B types), Controlled Oral Word Association test (COWA) Visuospatial function: Rey complex figure test Language: Short form of K-BNT Memory: The Korean version of the California Verbal Learning Test (KCVLT) for verbal memory and the Rey complex figure test of visual memory
Effects on sleepiness | 6th month
  Clinical questionnaire
  - Epworth Sleepiness Scale
Effects on seizures | 6th month
  Seizure frequency per month
Effects on depression | 6th month
  BDI (Beck Depression Index)

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Young Jung, M.D, Ph.D, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Ahn SJ, Kim TJ, Cha KS, Jun JS, Byun JI, Shin YW, Sunwoo JS, Lee S, Yu KS, Jang IJ, Chu K, Lee SK, Jung KY. Effects of perampanel on cognition and quantitative electroencephalography in patients with epilepsy. Epilepsy Behav. 2021 Feb;115:107514. doi: 10.1016/j.yebeh.2020.107514. Epub 2020 Dec 14. PMID 33328106